CLINICAL TRIAL: NCT05413980
Title: A Non-randomized, Non-Interventional, Prospective, Multicenter, Post Marketing Surveillance Study to Assess the Antibacterial Effectiveness and Safety of 0.5% Moxifloxacin Hydrochloride Ophthalmic Solution in Perioperative (Preoperative and Postoperative) Sterilization in Patients Undergoing Ophthalmic Surgery
Brief Title: Effectiveness and Safety of 0.5% Moxifloxacin Hydrochloride Ophthalmic Solution in Perioperative Sterilization in Patients Undergoing Ophthalmic Surgery
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CUKG489C1IN01
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Post Operative Endophthalmitis
Keywords: Moxifloxacin Hydrochloride Ophthalmic Solution; Ophthalmic Surgery; Antibacterial Effectiveness; NIS; India; preoperative; postoperative; endophthalmitis; perioperative sterilization; efficacy; safety
MeSH Terms: conditions — Endophthalmitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Moxifloxacin hydrochloride ophthalmic solution: patients prescribed with 0.5% Moxifloxacin hydrochloride ophthalmic solution during the perioperative (preoperative and postoperative) period of ophthalmic surgery.
  Interventions: Other: Moxifloxacin hydrochloride ophthalmic solution

INTERVENTIONS:
Other: Moxifloxacin hydrochloride ophthalmic solution — Prospective observational study. There is no treatment allocation. Patients prescribed with 0.5% Moxifloxacin hydrochloride ophthalmic solution during the perioperative period of ophthalmic surgery are eligible to enroll into this study.

SUMMARY:
This is a non-interventional, uncontrolled, prospective, multicenter, post marketing surveillance study.

DETAILED DESCRIPTION:
The study treatment i.e., 0.5% Moxifloxacin hydrochloride ophthalmic solution will be prescribed as per approved label; the assignment of the patient to the therapy will be decided within the current practice and the medical indication and will clearly be separated from the decision to include the patient in the study.

The treatment period for each patient will be maximum 17 days from start of Moxifloxacin treatment. Study visit will be 1 day prior to surgery, day of surgery (Day 0) and 1 (day of surgery / post surgery), 7, and 14 days post-op (Note: Since its non-interventional study, the eligibility confirmation can be 1 or 2 days prior to the surgery depending on investigator's discretion).

After the patients sign the informed consent, the patients will be advised to start with Moxifloxacin ophthalmic solutions 2 days prior to the surgery and will be advised to administer it 5 times a day. On the Day 0, day of the surgery, the patient will be instilled 1 drop of Moxifloxacin in the eye which will be operated prior to surgery and 1 drop twice post surgery. From Day 1 post surgery, patient will have 1 drop of Moxifloxacin instilled three times a day up to Day 14 (14 days after surgery). If there are any signs and symptoms of endophthalmitis, then at the investigator's discretion, Gram Stain & Culture assessment of aqueous & vitreous fluid may be performed post surgery on Days 1, 7, and 14.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years of age, who have been prescribed 0.5% Moxifloxacin drops preoperatively and postoperatively for 2 weeks after ocular Surgery
* Patient or legally acceptable representative (LAR) willing to voluntarily provide signed informed consent for participation in the study

Exclusion Criteria:

* Patients with known history of hypersensitivity to fluoroquinolones
* Patients with history of serious underlying ocular or systemic disease or complication before surgery
* Patients diagnosed with an extraocular bacterial, viral, fungal infection prior to surgery
* Patients who have been administered other topical antibacterial agents within 24 hours of Moxifloxacin administration or systemic antibacterial agents within 72 hours of Moxifloxacin administration
* Patients who have planned to undergo cataract surgery in both eyes on same day
* Patients who have participated in another clinical study within 30 days prior to the start of this study
* Pregnant women/lactating mothers/ women suspected to be pregnant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients that are to undergo ocular surgery and are to be treated with Moxifloxacin and have provided informed consent
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2024-01-27 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Post-op endophthalmitis rate up to Day 14 | Up to Day 14 after surgery
  The post-op endophthalmitis rate = (No of patients in whom endophthalmitis occurred in post-op period up to Day 14/ no of enrolled patients) X 100

SECONDARY OUTCOMES:
Number of patients with diagnosis of suspected endophthalmitis using microbiological culture and Gram stain of aqueous and vitreous fluids | Day 1, Day 7, Day 14 after surgery
  Number of patients with diagnosis of suspected endophthalmitis using microbiological culture and Gram stain of aqueous and vitreous fluids to be collected
Number of patients assessed for infection using 4 clinical signs post-surgery | Day 1, Day 7, Day 14 after surgery
  To assess for infection using 4 clinical signs post-surgery:
  1. Drop in vision
  2. Pain and redness
  3. Swelling
  4. Purulent discharge
  It will be recorded and measured as present or absent.
Number and proportion of patients with ocular adverse events (AEs) after surgery | Up to Day 16 after surgery
  Number and proportion of patients with ocular adverse events (AEs) after surgery to be collected

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- India (7):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Varanasi, Uttar Pradesh
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Delhi

IPD SHARING:
Plan to Share IPD: No